CLINICAL TRIAL: NCT04211311
Title: "Feasibility of High-intensity Interval Training (HIIT) as Hybrid Exercise Using Functional Electrical Stimulation Leg-cycling (FEScycling) and Ski Ergometer (SkiErg) With the Arms for People With Chronic Spinal Cord Injury Paraplegia"
Brief Title: Hybrid High-intensity Interval Training for Persons With Spinal Cord Injury. A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: d4qxwjy6
Record Dates: First submitted 2019-10-10; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES-legcycling with voluntary arm-work (Experimental): FES-legcycling combined with arm ski-ergometer or arm-cycling
  Interventions: Other: hybrid high-intensity training

INTERVENTIONS:
Other: hybrid high-intensity training — FES-legcycling combined with either arm skiergometer or arm-cycling in 4 x 4 min. intervals at 90% peak power output, 3 times a week for 8 weeks

SUMMARY:
This study examines safety and feasibility of a study protocol using a combination of functional electrical legcycling with voluntary armwork (hybrid training) as either skiergometer or armcycling in high intensity intervals for persons with spinal cord injury paraplegia.

DETAILED DESCRIPTION:
Cardiovascular disease is one of the most common causes of early death in people with spinal cord injury. Physical activity at high intensity is known to reduce the risk of cardiovascular disease in other patient groups.

During aerobic training, combining functional electrical stimulation (FES) with voluntary arm-work induces a higher oxygen uptake than FES cycling alone and high intensity interval training induces higher oxygen uptake than training at continuous intensity. The hypothesis is that combining hybrid training with high-intensity induces even higher oxygen uptake thereby reducing the risk of cardiovascular disease. This training modality has not been tested before, so before conducting a randomized controlled trial testing the effect of this training modality on oxygen uptake, the aim was to asses safety and feasibility of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury paraplegia,
* complete and incomplete lesions,
* ability to be electrically stimulated,
* willing to train 3 times a week at high intensity

Exclusion Criteria:

* heart pacemaker or other heart problems contradicting high intensity aerobic training,
* pregnancy,
* unstable fractures,
* cancer,
* heterotopic ossification,
* myositis ossificans,
* severe osteoporosis,
* pressure ulcers,
* newly implanted metal,
* newly surgery,
* frequent episodes of autonomic hyperreflexia,
* very high or low blood pressure,
* dislocation or subluxation of joints
* high level of shoulder pain at study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events | 8 weeks
  Assessed by number of incidences of autonomic hyperreflexia or acute cardiac events
Shoulder pain | 8 weeks
  Measured using Wheelchair Shoulder Pain Index (WUSPI), a 15 item questionnaire measuring shoulder pain during daily activities. Each item is scored on a 10 mm visual analog scale with anchors no pain to worst pain ever. Total index score range from 0 - 100. Within each item there is a not applicable option. The score used is performance corrected WUSPI score, dividing total index score by number of item responses and multiplied by 15. Higher score indicate higher level of shoulder pain.
compliance | 8 weeks
  Assessed with number of dropouts and proportion of fulfilled training minutes
intensity | 8 weeks
  Assessed as mean intensity of the 4 x 4 min. intervals as proportion of peak watt measured at baseline test. Peakwatt for FES-cycling was defined as an average of the three highest watt values within 30 sec. For skiergometer peak watt was defined as the highest average of one min. splits.

SECONDARY OUTCOMES:
Peak oxygen uptake | 8 weeks
  Assessed measuring pulmonary gas exchange. Peak oxygen uptake is defined as respiratory exchange ratio of 1.05 or higher, concentration of blood lactate of 7 mmol/l or more and subjective rating of perceived exertion on the Borg 6-20 scale of min. 16.
leisure time physical activity | 8 weeks
  leisure time physical activity measured with leisure time physical activity questionnaire - SCI (LTPAQ-SCI), asking number of min. spent performing low-, moderate and high intensity leisure time physical activity pr. day, scored by multiplying number of min by number of days yielding number of minutes of leisure time physical activity per week.
health related quality of life | 8 weeks
  health related quality of life measured with Short Form 36 (SF-36), categorically based on a three to six categories Likert scale. An algorithm transforms the scores into a 0-100 scoring system, with higher scores indicating better quality of life
Fatigue | 8 weeks
  Assessed with the Multi Dimensional Fatigue Inventory (MFI-20) covering 5 dimensions of fatigue which are scored using a five level scale. Sub scale scores range 4-20 are calculated as the sum of item ratings and total fatigue score range 20-100 is calculated as the sum of sub scale scores with higher scores indicating lower level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Juul-Kristensen, Assoc Prof, Study Director — Denmark, University of Southern Denmark, Odense, Funen, Denmark, 5230
Locations (1):
- Specialhospitalet for Polio og Ulykkesramte, Rødovre Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
No, due to the small sample size (8) as a feasibility study is, and the group is heterogeneous.

REFERENCES:
- [Derived] Vestergaard M, Jensen K, Juul-Kristensen B. Hybrid high-intensity interval training using functional electrical stimulation leg cycling and arm ski ergometer for people with spinal cord injuries: a feasibility study. Pilot Feasibility Stud. 2022 Feb 22;8(1):43. doi: 10.1186/s40814-022-00997-2. PMID 35193705